CLINICAL TRIAL: NCT00969956
Title: Time to Complications Occurs in Diabetes. Risk Factors Determine When Diabetes Complications Occur
Brief Title: Time To Complications Occurs in Diabetes
Status: Terminated | Type: Observational
Why Stopped: Local regulations
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mats Bonnier, MD, Karolinska Institutet
Other Study IDs: TTCOD
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Retinopathy; Nephropathy; Diabetic Neuropathy; Vascular Disease; Ischemic Heart Disease
Keywords: Diabetes, Complication, Cardio-vascular disease
MeSH Terms: conditions — Retinal Diseases; Kidney Diseases; Diabetic Neuropathies; Vascular Diseases; Myocardial Ischemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: 150 Type 1 Diabetes, duration of 15 years (+/- 2 years) and 150 Type 2 Diabetes, duration of 2 years (+/- 2 years) (50% women / men)
- Group B: 150 Type 1 Diabetes, duration of 20 years (+/- 2 years) and 150 Type 2 Diabetes, duration of 7 years (+/- 2 years) (50% women / men)
- Group C: 150 Type 1 Diabetes, duration of 25 years (+/- 2 years) and 150 Type 2 Diabetes duration of 12 years (+/- 2 years) (50% women / men)
- Group D: 50 LADA (Late Autoimmune Diabetes in Adults), debut after 35 years of age, duration of 5-10 years (50% women / men)

SUMMARY:
Diabetes causing serious complications is well known. In this study the aim is to follow 950 patients with diabetes for 15 years to study when, in who and how the diabetes complications occurs.

DETAILED DESCRIPTION:
Background:

That diabetes cause serious diabetic complications from the eyes, kidneys, nerves and large vessels is known. Good metabolic control during the first 8-10 years has been shown to delay and even alleviate diabetes complications, but not entirely prevent them. When complications occur early after diabetes onset there are also likely genetic causes. If the various diabetes complications have different formation mechanisms or different sensitivity of blood sugar impact is not studied previously.

Hypothesis:

1. Genetic factors determine increased risk of early onset of complications.
2. Oxidative stress increases the risk of complications.
3. Inflammation, hyperlipidemia and hypertension leads to hypoxia and oxidative stress.
4. Combined hypoxia and hyperglycemia leads to complications.

Questionnaires:

1. Are there measurable risk factors that indicate different sensitivity to develop diabetes complications?
2. Are there differences between men and women?
3. Are there differences between type 1 and type 2 diabetes?

Knowledge achievements:

Being able to anticipate and prevent diabetes complications with specific approaches would mean major benefits for patients and society.

Inclusions criteria:

Diabetes type 1, 2 or LADA: 18-75 years of age. Group A: 150 Type 1 Diabetes, duration 15 years (+/- 2 years) and 150 Type 2 Diabetes 2 years (+/- 2 years) (50% K / M) Group B: 150 Type 1 Diabetes, duration 20 years (+/- 2 years) and 150 Type 2 Diabetes 7 years (+/- 2 years) (50% K / M) Group C: 150 Type 1 Diabetes, duration 25 years (+/- 2 years) and 150 Type 2 Diabetes 12 years (+/- 2 years) (50% K / M) Group D: 50 LADA, onset after 35 years of age, duration of 5-10 years (50% K / M)

Follow-up visits:

Group A: After 3, 8 and 13 years Group B: After 5, 10 and 15 years Group C: After 5, 10 and 15 years Group D: After 3, 8 and 13 years

Definitions:

Type 1 Diabetes: Positive ICA-antibodies and/or GAD-antibodies and/or neg C-peptide. Debut <30 years of age.

Type 2 Diabetes: Negative ICA-antibodies and GAD-antibodies and pos C-peptide (> 0.35 mmol/l).

LADA: Positive ICA-antibodies and/or GAD-antibodies. Debut >35 years of age.

Retinopathy: Level of retinopathy based on fundus photography judged by experienced ophthalmologist and classified according to DRP classification in five steps: 1. No retinopathy, 2. Mild non-proliferative retinopathy, 3. Moderate non-proliferative retinopathy, 4. Severe non-proliferative retinopathy, 5. Proliferative retinopathy

ESRD (end stage renal disease): Dialysis or transplantation demanding, GFR (glomerular filtration rate) <10 ml/min.

Overt nephropathy: Albumin excretion at least two consecutive measurements,≥ 300 mg/L and/or S-Creatinine > 100 women and > 110 mmol/l in men.

Incipient nephropathy: Albuminuria between 30 - 300mg/L or Urine albumin/Creatinine >3.

Hypertension: Measured blood pressure in sitting position after 10 minutes rest, at least two consecutive measurements with at least 4 weeks in between, ≥ 130/80.

Hyperlipidemia: ApoA-1/ApoB: >0.5 and/or Triglycerides >1,7 mmol/L and/or LDL >2.5 mmol/L and/or HDL women <1.3, men <1.1 mmol/L and/or cholesterol >4.5 mmol/L.

Heart disease: History of myocardial infarction, angina pectoris and/or ischemic heart disease (file noted). Pharmacological treatment for ischemic heart disease, heart failure or pathological electrocardiographic changes according to Minnesota code.

Cerebrovascular disease: Deemed to have been: if recorded in the patients file and/or if pathological findings demonstrated on CT/MR.

Peripheral vascular disease: Ankle Index <0.9 (blood pressure arm>ankle) Clinical macroangiopathy, (absence of peripheral pulse) or history typical for claudication intermittens.

Neuropathy: Foot investigation: According to international consensus for the investigation and risk assessment of diabetic feet with a view of peripheral autonomic neuropathy (PAN) and peripheral sensory neuropathy (PSN).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1, 2 or LADA: 18-75 years of age.
* Group A: 150 Type 1 Diabetes, duration 15 years (+/-2 years) and 150 Type 2
* Diabetes 2 years (+/-2 years) (50% F/M)
* Group B: 150 Type 1 Diabetes, duration 20 years (+/-2 years) and 150 Type 2
* Diabetes 7 years (+/-2 years) (50% F/M)
* Group C: 150 Type 1 Diabetes, duration 25 years (+/-2 years) and 150 Type 2
* Diabetes 12 years (+/-2 years) (50% F/M)
* Group D: 50 LADA, onset after 35 years of age, duration of 5-10 years (50% F/M)
* Type 1 Diabetes: Positive ICA antibodies and/or GAD-antibodies and/or neg C-peptide. Debut <30 years of age.
* Type 2 Diabetes: Negative ICA-antibodies and GAD-antibodies and pos C-peptide (>0.35 mmol/l).
* LADA: Positive ICA-antibodies and/or GAD-antibodies. Debut >35 years of age.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Typ 1, Typ 2 and LADA Diabetics from the diabetic clinic at Sophiahemmet, Stockholm, Sweden
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Time to nephropathy | 0, 3-5, 8-10 and 13-15 years
Time to autonomous neuropathic ulcers and Amputation | 0, 3-5, 8-10 and 13-15 years
Time to peripheral neuropathy | 0, 3-5, 8-10 and 13-15 years
Time to peripheral Macro-Vascular Disease, chronic Foot ulcers and Amputation | 0, 3-5, 8-10 and 13-15 years
Time to retinopathy | 0, 3-5, 8-10 and 13-15 years

SECONDARY OUTCOMES:
DNA | 0, 3-5, 8-10 and 13-15 years
Endothelial markers | 0, 3-5, 8-10 and 13-15 years
Blood lipids | 0, 3-5, 8-10 and 13-15 years
CRP | 0, 3-5, 8-10 and 13-15 years
Oxidative stress | 0, 3-5, 8-10 and 13-15 years
Q10 | 0, 3-5, 8-10 and 13-15 years
IGFBP-1 | 0, 3-5, 8-10 and 13-15 years
IGF-1 | 0, 3-5, 8-10 and 13-15 years
Inflammatory markers | 0, 3-5, 8-10 and 13-15 years
Seated blood pressure | 0, 3-5, 8-10 and 13-15 years
Pulse | 0, 3-5, 8-10 and 13-15 years
Weight | 0, 3-5, 8-10 and 13-15 years
BMI | 0, 3-5, 8-10 and 13-15 years
Waistlines | 0, 3-5, 8-10 and 13-15 years

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Brismar, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Molecular Medicine and Surgery, Rolf Luft Research centre for Diabetes and Endocrinology, Stockholm, Sweden

REFERENCES:
- [Background] Gaede P, Pedersen O. Intensive integrated therapy of type 2 diabetes: implications for long-term prognosis. Diabetes. 2004 Dec;53 Suppl 3:S39-47. doi: 10.2337/diabetes.53.suppl_3.s39. PMID 15561920
- [Background] Genuth S. Insights from the diabetes control and complications trial/epidemiology of diabetes interventions and complications study on the use of intensive glycemic treatment to reduce the risk of complications of type 1 diabetes. Endocr Pract. 2006 Jan-Feb;12 Suppl 1:34-41. doi: 10.4158/EP.12.S1.34. PMID 16627378
- [Background] Hadi HA, Suwaidi JA. Endothelial dysfunction in diabetes mellitus. Vasc Health Risk Manag. 2007;3(6):853-76. PMID 18200806
- [Background] Brismar K, Fernqvist-Forbes E, Wahren J, Hall K. Effect of insulin on the hepatic production of insulin-like growth factor-binding protein-1 (IGFBP-1), IGFBP-3, and IGF-I in insulin-dependent diabetes. J Clin Endocrinol Metab. 1994 Sep;79(3):872-8. doi: 10.1210/jcem.79.3.7521354.
- [Background] Penckofer S, Kouba J, Wallis DE, Emanuele MA. Vitamin D and diabetes: let the sunshine in. Diabetes Educ. 2008 Nov-Dec;34(6):939-40, 942, 944 passim. doi: 10.1177/0145721708326764. PMID 19075078
- [Background] Vinik AI, Maser RE, Mitchell BD, Freeman R. Diabetic autonomic neuropathy. Diabetes Care. 2003 May;26(5):1553-79. doi: 10.2337/diacare.26.5.1553. PMID 12716821
- [Background] Kotronen A, Lewitt M, Hall K, Brismar K, Yki-Jarvinen H. Insulin-like growth factor binding protein 1 as a novel specific marker of hepatic insulin sensitivity. J Clin Endocrinol Metab. 2008 Dec;93(12):4867-72. doi: 10.1210/jc.2008-1245. Epub 2008 Sep 16. PMID 18796514
- [Background] King GL. The role of inflammatory cytokines in diabetes and its complications. J Periodontol. 2008 Aug;79(8 Suppl):1527-34. doi: 10.1902/jop.2008.080246. PMID 18673007
- [Background] Pop-Busui R. Cardiac autonomic neuropathy in diabetes: a clinical perspective. Diabetes Care. 2010 Feb;33(2):434-41. doi: 10.2337/dc09-1294. No abstract available. PMID 20103559
- [Background] Pickup JC. Inflammation and activated innate immunity in the pathogenesis of type 2 diabetes. Diabetes Care. 2004 Mar;27(3):813-23. doi: 10.2337/diacare.27.3.813. PMID 14988310
- [Background] Gomes F, Telo DF, Souza HP, Nicolau JC, Halpern A, Serrano CV Jr. Obesity and coronary artery disease: role of vascular inflammation. Arq Bras Cardiol. 2010 Feb;94(2):255-61, 273-9, 260-6. doi: 10.1590/s0066-782x2010000200021. English, Portuguese, Spanish. PMID 20428625
- [Background] Arai Y, Kojima T, Takayama M, Hirose N. The metabolic syndrome, IGF-1, and insulin action. Mol Cell Endocrinol. 2009 Feb 5;299(1):124-8. doi: 10.1016/j.mce.2008.07.002. Epub 2008 Jul 11. PMID 18672019
- [Background] Eriksson A, Attvall S, Bonnier M, Eriksson JW, Rosander B, Karlsson FA. Short-term effects of metformin in type 2 diabetes. Diabetes Obes Metab. 2007 Jul;9(4):483-9. doi: 10.1111/j.1463-1326.2006.00624.x. PMID 17587390
- [Background] Galic S, Oakhill JS, Steinberg GR. Adipose tissue as an endocrine organ. Mol Cell Endocrinol. 2010 Mar 25;316(2):129-39. doi: 10.1016/j.mce.2009.08.018. Epub 2009 Aug 31. PMID 19723556
- [Background] Salpeter SR, Buckley NS, Kahn JA, Salpeter EE. Meta-analysis: metformin treatment in persons at risk for diabetes mellitus. Am J Med. 2008 Feb;121(2):149-157.e2. doi: 10.1016/j.amjmed.2007.09.016. PMID 18261504
- [Background] Orchard TJ, Temprosa M, Goldberg R, Haffner S, Ratner R, Marcovina S, Fowler S; Diabetes Prevention Program Research Group. The effect of metformin and intensive lifestyle intervention on the metabolic syndrome: the Diabetes Prevention Program randomized trial. Ann Intern Med. 2005 Apr 19;142(8):611-9. doi: 10.7326/0003-4819-142-8-200504190-00009. PMID 15838067
- [Background] Alagona P Jr. Beyond LDL cholesterol: the role of elevated triglycerides and low HDL cholesterol in residual CVD risk remaining after statin therapy. Am J Manag Care. 2009 Mar;15(3 Suppl):S65-73. PMID 19355805
- [Background] Hemmingsen B, Lund SS, Gluud C, Vaag A, Almdal TP, Hemmingsen C, Wetterslev J. Targeting intensive glycaemic control versus targeting conventional glycaemic control for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2013 Nov 11;(11):CD008143. doi: 10.1002/14651858.CD008143.pub3. PMID 24214280
- [Background] Fullerton B, Jeitler K, Seitz M, Horvath K, Berghold A, Siebenhofer A. Intensive glucose control versus conventional glucose control for type 1 diabetes mellitus. Cochrane Database Syst Rev. 2014 Feb 14;2014(2):CD009122. doi: 10.1002/14651858.CD009122.pub2. PMID 24526393